CLINICAL TRIAL: NCT03137953
Title: Role of Imaging to Predict the Deep Surgical Margin in Gingivobuccal Complex Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HealthCare Global Enterprise Ltd. (Industry)
Responsible Party: Principal Investigator, Vishal U S Rao, Senior Consultant, HealthCare Global Enterprise Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HCG/SX/002/2016
Record Dates: First submitted 2017-02-13; First posted 2017-05-03 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Buccal Mucosa Cancer; Gingival Cancer
MeSH Terms: interventions — Postmortem Imaging

STUDY DESIGN:
Intervention Model Description: Examination of the distance between the skin and the base of the tumour would be evaluated clinically (skin Pinch Test) and by CT/MRI with contrast. Post resection, histopathological examination of tumour margins would confirm if the base of the tumour is free or not. The proportion of cases where skin is preserved would be compared to the proportion of cases where skin would have been preserved based on clinical examination would be assessed.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clinical and Imaging (Experimental): Subjects in this arm would undergo clinical evaluation of skin involvement followed by Radiological Imaging (CT/MRI) based evaluation of the distance between the base of the tumor and the skin. Based on this distance, the skin would either be conserved or not during tumor resection.
  Interventions: Procedure: Clinical Evaluation; Diagnostic Test: Radiological Imaging

INTERVENTIONS:
Procedure: Clinical Evaluation — The skin pinch test would be done by three independent oncologists to assess ability for skin conservation. The decision for skin conservation would be taken by the surgeon intra-operatively based on clinical and radiological assessments.
Diagnostic Test: Radiological Imaging — Computed Tomography or Magnetic Resonance Imaging would be done by a radiologist and used to measure the distance between tumor and skin which would guide the decision for skin presevation. The decision for skin conservation would be taken by the surgeon intra-operatively based on clinical and radiological assessments.

SUMMARY:
In gingivobuccal complex tumors, the skin margin is assessed by palpation (skin pinch test). There is no objective method of assessment of skin margin. This study is to evaluate the role of computed tomography/MRI with contrast in assessing the deep surgical margin.

DETAILED DESCRIPTION:
The patients of buccal mucosa squamous cell carcinomas after histopathological confirmation are selected for the study. As a routine computed tomography imaging/MRI with contrast will be done preoperatively.

The involvement of the skin is assessed by the palpation (skin pinch test). In imaging, the distance between the base of the tumour and the skin of the cheek is measured. If the distance between the base of the tumour and the skin is more than 5mm, then the skin is spared and the tumour is excised with 5 mm margin, if the distance is less than 5mm, then the skin is excised along with the tumour. The specimen will be sent for histopathological examination, and the depth of invasion of the tumour is measured and the clearance of the deep surgical margin is assessed.

The difference between clinical examination and imaging and histopathological confirmation of the specimen in determining the number of cases where skin preservation is done is assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients of buccal mucosa squamous cell carcinomas of stage 1,2 and 3 are included in the study
* Patient of all age groups are included in the study
* Both males and females are included in the study

Exclusion Criteria:

* Patients with buccal mucosa carcinomas, in whom the tumour is involving/fungating through the skin.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-06-30 (Estimated); Study Completion 2017-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients undergoing skin preservation surgeries | Data would be obtained on the day of Surgery
  Proportion of subjects who are to undergo skin preservation surgeries

CONTACTS AND LOCATIONS:
Overall Officials: Vishal US Rao, MS, Principal Investigator — Dept of Head & Neck Surgery, HealthCare Global Enterprises Ltd.
Locations (1):
- HealthCare Global Enterprises Ltd, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ota Y, Aoki T, Karakida K, Otsuru M, Kurabayashi H, Sasaki M, Nakamura N, Kajiwara H. Determination of deep surgical margin based on anatomical architecture for local control of squamous cell carcinoma of the buccal mucosa. Oral Oncol. 2009 Jul;45(7):605-9. doi: 10.1016/j.oraloncology.2008.08.010. Epub 2008 Nov 20. PMID 19026588
- [Background] Liao CT, Wang HM, Ng SH, Yen TC, Lee LY, Hsueh C, Wei FC, Chen IH, Kang CJ, Huang SF, Chang JT. Good tumor control and survivals of squamous cell carcinoma of buccal mucosa treated with radical surgery with or without neck dissection in Taiwan. Oral Oncol. 2006 Sep;42(8):800-9. doi: 10.1016/j.oraloncology.2005.11.020. Epub 2006 Feb 2. PMID 16458038
- [Background] Coppen C, de Wilde PC, Pop LA, van den Hoogen FJ, Merkx MA. Treatment results of patients with a squamous cell carcinoma of the buccal mucosa. Oral Oncol. 2006 Sep;42(8):795-9. doi: 10.1016/j.oraloncology.2005.11.017. Epub 2006 Mar 10. PMID 16529979